CLINICAL TRIAL: NCT00000739
Title: Comparison of Two Dosage Regimens of Oral Dapsone for Prophylaxis of Pneumocystis Carinii Pneumonia in Pediatric HIV Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Jacobus Pharmaceutical (Industry)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 179; 11154 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: Pneumonia, Pneumocystis Carinii; HIV Infections
Keywords: Pneumonia, Pneumocystis carinii; Dapsone; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Drug Administration Schedule
MeSH Terms: conditions — Pneumonia, Pneumocystis; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Dapsone

INTERVENTIONS:
Drug: Dapsone

SUMMARY:
Primary: To compare the toxicity of daily versus weekly dapsone in HIV-infected infants and children; to study the pharmacokinetics of orally administered dapsone in HIV-infected infants and children.

Secondary: To obtain information on the rate of Pneumocystis carinii pneumonia ( PCP ) breakthrough in children receiving two different dose regimens of dapsone.

Prophylaxis for Pneumocystis carinii pneumonia ( PCP ) is recommended for all HIV-infected children considered to be at high risk. Approximately 15 percent of children are intolerant to trimethoprim / sulfamethoxazole, the first choice drug for PCP prophylaxis. Since many children are also unable to take or tolerate aerosolized pentamidine, dapsone is a second choice for PCP prophylaxis. The most favorable dose regimen for dapsone has not been established.

DETAILED DESCRIPTION:
Prophylaxis for Pneumocystis carinii pneumonia ( PCP ) is recommended for all HIV-infected children considered to be at high risk. Approximately 15 percent of children are intolerant to trimethoprim / sulfamethoxazole, the first choice drug for PCP prophylaxis. Since many children are also unable to take or tolerate aerosolized pentamidine, dapsone is a second choice for PCP prophylaxis. The most favorable dose regimen for dapsone has not been established.

Ninety-six HIV-infected infants and children who are intolerant to trimethoprim / sulfamethoxazole ( TMP / SMX ) are randomized to receive oral dapsone in a lower dose once daily or at a higher dose once weekly. Treatment continues until the last patient enrolled has received at least 3 months of therapy. Blood samples are drawn between weeks 4 and 8, at weeks 12 and 24, and every 3 months thereafter during dapsone administration.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Rifampin and rifampin derivatives for up to 1 week during the study.
* Rifabutin or other drugs that could alter dapsone metabolism (if prescribed by the child's primary care physician).

Patients must have:

* Evidence of HIV infection.

PER AMENDMENT 11/16/95:

* Children who require prophylaxis. (Was written - Risk of developing PCP.)
* Known intolerance to TMP / SMX.
* Consent of parent or guardian. Patients entering this study may be co-enrolled in other ACTG pediatric studies.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Glucose-6-phosphate dehydrogenase deficiency.
* Known allergy to dapsone.

Concurrent Medication:

Excluded:

* Rifampin, rifampin derivatives, or oxidant drugs for more than 1 week.

Patients with the following prior conditions are excluded:

* Serious or life-threatening reactions to TMP / SMX (e.g., anaphylaxis, Stevens-Johnson syndrome, hypotension) that would contraindicate therapy with sulfa drugs.

Prior Medication:

Excluded:

* Prior dapsone.
* Rifampin, rifampin derivatives, or oxidant drugs within 1 week prior to study entry.
* TMP / SMX within 7 days prior to study entry (and toxicity must be clearly resolving).

Prior Treatment:

Excluded:

* RBC transfusion within 4 weeks prior to study entry.

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96
Dates: Study Completion 1998-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: McIntosh K, Study Chair; Cooper E, Study Chair
Locations (46):
- United States (43):
  - Long Beach Memorial Med. Ctr., Miller Children's Hosp., Long Beach, California
  - Usc La Nichd Crs, Los Angeles, California
  - UCLA-Los Angeles/Brazil AIDS Consortium (LABAC) CRS, Los Angeles, California
  - Children's Hosp. & Research Ctr. Oakland, Ped. Clinical Research Ctr. & Research Lab., Oakland, California
  - UCSD Maternal, Child, and Adolescent HIV CRS, San Diego, California
  - Harbor - UCLA Med. Ctr. - Dept. of Peds., Div. of Infectious Diseases, Torrance, California
  - Univ. of Colorado Denver NICHD CRS, Aurora, Colorado
  - Children's National Med. Ctr., ACTU, Washington D.C., District of Columbia
  - Howard Univ. Washington DC NICHD CRS, Washington D.C., District of Columbia
  - Univ. of Florida Jacksonville NICHD CRS, Jacksonville, Florida
  - Univ. of Miami Ped. Perinatal HIV/AIDS CRS, Miami, Florida
  - Emory Univ. School of Medicine, Dept. of Peds., Div. of Infectious Diseases, Atlanta, Georgia
  - Cook County Hosp., Chicago, Illinois
  - Chicago Children's CRS, Chicago, Illinois
  - Univ. of Chicago - Dept. of Peds., Div. of Infectious Disease, Chicago, Illinois
  - Univ. of Illinois College of Medicine at Chicago, Dept. of Peds, Chicago, Illinois
  - Tulane/LSU Maternal/Child CRS, New Orleans, Louisiana
  - HMS - Children's Hosp. Boston, Div. of Infectious Diseases, Boston, Massachusetts
  - BMC, Div. of Ped Infectious Diseases, Boston, Massachusetts
  - Baystate Health, Baystate Med. Ctr., Springfield, Massachusetts
  - WNE Maternal Pediatric Adolescent AIDS CRS, Worcester, Massachusetts
  - Children's Hospital of Michigan NICHD CRS, Detroit, Michigan
  - UMDNJ - Robert Wood Johnson, New Brunswick, New Jersey
  - St. Joseph's Hosp. & Med. Ctr. of New Jersey, Paterson, New Jersey
  - SUNY Downstate Med. Ctr., Children's Hosp. at Downstate NICHD CRS, Brooklyn, New York
  - North Shore-Long Island Jewish Health System, Dept. of Peds., Great Neck, New York
  - Schneider Children's Hosp., Div. of Infectious Diseases, New Hyde Park, New York
  - NYU Med. Ctr., Dept. of Medicine, New York, New York
  - Columbia IMPAACT CRS, New York, New York
  - Incarnation Children's Ctr., New York, New York
  - Harlem Hosp. Ctr. NY NICHD CRS, New York, New York
  - Univ. of Rochester ACTG CRS, Rochester, New York
  - Strong Memorial Hospital Rochester NY NICHD CRS, Rochester, New York
  - SUNY Stony Brook NICHD CRS, Stony Brook, New York
  - SUNY Upstate Med. Univ., Dept. of Peds., Syracuse, New York
  - DUMC Ped. CRS, Durham, North Carolina
  - Case CRS, Cleveland, Ohio
  - The Children's Hosp. of Philadelphia IMPAACT CRS, Philadelphia, Pennsylvania
  - St. Christopher's Hosp. for Children, Philadelphia, Pennsylvania
  - Med. Univ. of South Carolina, Div. of Ped. Infectious Diseases, Charleston, South Carolina
  - St. Jude/UTHSC CRS, Memphis, Tennessee
  - Childrens Hosp. of the Kings Daughters, Norfolk, Virginia
  - UW School of Medicine - CHRMC, Seattle, Washington
- Puerto Rico (3):
  - Univ. Hosp. Ramón Ruiz Arnau, Dept. of Peds, Bayamón
  - San Juan City Hosp. PR NICHD CRS, San Juan
  - Univ. of Puerto Rico Ped. HIV/AIDS Research Program CRS, San Juan

REFERENCES:
- [Background] Mirochnick M, Cooper E, McIntosh K. Pharmacokinetics of daily and weekly dapsone in HIV-infected children. Conf Retroviruses Opportunistic Infect. 1996 Jan 28-Feb 1;3rd:159
- [Background] Mirochnick M, Cooper E, Mcintosh K. Pharmacokinetics of daily and weekly dapsone in HIV-infected children. ACTG Protocol 179 Team. American Pediatric Association and Society for Pediatric Research annual meeting; 1996 May 6-10; Washington, D.C. Pediatr AIDS HIV Infect. 1996 Aug;7(4):280 (unnumbered abstract)
- [Background] Perrier M, Schwarz T, Gonzalez O, Brounts S. Squamous cell carcinoma invading the right temporomandibular joint in a Belgian mare. Can Vet J. 2010 Aug;51(8):885-7. PMID 21037891
- [Background] McIntosh K, Cooper E, Xu J, Mirochnick M, Lindsey J, Jacobus D, Mofenson L, Yogev R, Spector SA, Sullivan JL, Sacks H, Kovacs A, Nachman S, Sleasman J, Bonagura V, McNamara J. Toxicity and efficacy of daily vs. weekly dapsone for prevention of Pneumocystis carinii pneumonia in children infected with human immunodeficiency virus. ACTG 179 Study Team. AIDS Clinical Trials Group. Pediatr Infect Dis J. 1999 May;18(5):432-9. doi: 10.1097/00006454-199905000-00007. PMID 10353516